CLINICAL TRIAL: NCT00411489
Title: Use of a New Endosurgical Operating System for Endoscopic Stoma and Pouch Reduction in Patients With Weight Regain Following Roux-En-Y Bypass Surgery
Brief Title: Endoscopic Stomach and Pouch Reduction in Patients With Weight Regain Following Roux-En-Y Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USGI Medical (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: TP0165; TP0165
Record Dates: First submitted 2006-12-12; First posted 2006-12-14 (Estimated); Last update posted 2008-03-18 (Estimated); Status verified 2007-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

INTERVENTIONS:
Procedure: endolumenal surgery

SUMMARY:
The Roux-En-Y gastric bypass procedure is the most commonly performed bariatric procedure in the United States. Despite initial weight loss, some patients experience weight regain that may be related to an increase in the size of the gastric pouch and/or stoma. A second surgical procedure to reduce the size of the pouch and/or stoma is typically associated with a higher risk of death or complications than the original gastric bypass procedure. This study will evaluate a less invasive, endolumenal alternative to pouch and stoma revision as a means of producing weight loss in patients who have regained weight following gastric bypass.

ELIGIBILITY:
Inclusion Criteria:

* 18 yrs of age or older and < 65 yrs of age
* At least 2 yrs post-Roux-En-Y gastric bypass surgery
* Initially achieved at least 50% weight loss
* At enrollment, has regain at least 15% of weight loss
* BMI 40 or greater or 35 or greater with one or more co-morbidities
* Stoma diameter at least 20 mm
* Completes successful nutritional screening
* Is a candidate for a surgical revision procedure
* Is a reasonable risk to undergo general anesthesia
* Completes successful cardiopulmonary evaluation
* ASA Classification of less than or equal to III
* Able to provide written consent
* Able to return for protocol-specified evaluations

Exclusion Criteria:

* Esophageal stricture or other anatomy/condition that precludes passage of endolumenal instruments
* Previous bariatric revision procedure
* Has another causal factor for weight regain other than stoma or pouch dilatation
* Non-mobile or has significant impairment of mobility that will limit compliance with post-op exercise program

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

PRIMARY OUTCOMES:
weight loss

CONTACTS AND LOCATIONS:
Overall Officials: Lee L Swanstrom, MD, Principal Investigator — Oregon Clinic
Locations (4):
- United States (4):
  - Lahey Clinic, Burlington, Massachusetts
  - Mt. Sinai School of Medicine, New York, New York
  - Columbia-Presbyterian Medical Center, New York, New York
  - Oregon Clinic, Portland, Oregon